CLINICAL TRIAL: NCT04546308
Title: Central Blood Pressure and Arterial Hemodynamic Responses to High-intensity Resistance Exercise Training - the Application of Ultrafast Ultrasound Analysis
Brief Title: Central Arterial Hemodynamics and Resistance Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 201903034RIND
Record Dates: First submitted 2020-09-06; First posted 2020-09-14 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-02

CONDITIONS: Hypertension; Cardiovascular Risk Factor
Keywords: Exercise; Ultrafast ultrasound
MeSH Terms: conditions — Hypertension; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise training (Experimental): The participants will undergo 8 weeks of whole-body resistance exercise training followed by a 4-week detraining. The central hemodynamic and muscle stiffness variables will be measured pre, post-training, and post-detraining.
  Interventions: Other: Resistance exercise training
- Sedentary control (No Intervention): The participants will undergo 12 weeks of intervention without exercise training. The central hemodynamic and muscle stiffness variables will be measured pre, 8th, and 12th week.

INTERVENTIONS:
Other: Resistance exercise training — Eight weeks whole-body resistance exercise training (80%1 repetition maximal, 3 sessions per week) followed by a 4-week detraining intervention
  Arms: Exercise training

SUMMARY:
Resistance exercise training is one of the popular exercise modes that has been drawn the public's attention. However, existing evidence showed high-intensity resistance exercise training-induced negative adaptation on vascular function and blood pressure responses. Upper-body resistance exercise training is more likely to induced arterial stiffening, which has been shown to be gender-dependent. It is still unknown whether age also plays a role. We like to test the hypothesis that high-intensity upper body resistance exercise may lead to a higher increase of arterial stiffness, central blood pressure, and hemodynamic parameters in younger adults than older adults. We also hypothesize high intensity resistance training could contribute to greater central hemodynamic responses and muscle stiffness than the control; the change of muscle stiffness correlates with the change of hemodynamic parameters. Collectively, study 1 in this project is aimed to recruit 40 apparently healthy young (20-35yrs) and middle-aged to older adults (50-75yrs) into this study followed by upper-body or lower-body high-intensity exercise (80% 1 repetition maximum, 10 reps, 4 sets) by a randomized order. Blood draw, central blood pressure, hemodynamics will be performed and obtained at pre-, immediately-post, 20min, 40mins, and 60 mins post-exercise. Study 2 is aimed to investigate the effects of 8-week whole-body resistance exercise training followed by a 4-week detraining on above-measured variables in order to determine the long-term effects on resistance training. We will employee state-of-art ultrafast ultrasound to obtain muscle stiffness and carotid local pulse wave velocity. Endothelin-1 and catecholamines will also be measured to discover its underlying mechanisms on such stiffening effects induced by high-intensity resistance exercise.

ELIGIBILITY:
Inclusion Criteria:

* Healthy middle-aged to older adults

Exclusion Criteria:

* (1)BMI≧27, (2) Smoking habits for more than six months in the past, (3) Hypertension (blood pressure>140/90 mmHg), (4) Personal diabetes history (fasting blood sugar >126 mg /dL), heart disease, or other cardiovascular diseases, (5) bone damage, (6) regular use of supplements or vitamins

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-12-21 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Central blood pressure | Pre, 8th and 12th week
  Carotid blood pressure obtained by using tonometer
Muscle shear wave velocity | Pre, 8th and 12th week
  Shear wave velocity measured by using ultrafast ultrasound
Arterial pulse wave velocity | Pre, 8th and 12th week
  Pulse wave velocity measured by using a commercialized vascular monitor.

SECONDARY OUTCOMES:
Vascular related biomarkers | Pre, 8th and 12th week
  Catecholamines, endothelin-1

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No